CLINICAL TRIAL: NCT03653260
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety in Chinese Children
Brief Title: A Study to Evaluate the Efficacy and Safety of Zingo in Chinese Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: Zhaoke (Hefei) Pharmaceutical Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-ZK-007
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Catheter Site Pain; Pain, Acute; Anesthesia, Local
MeSH Terms: conditions — Acute Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Zingo) (Experimental): 0.5mg lidocaine at 20 bar pressure
  Interventions: Drug: Lidocaine (Zingo)
- Placebo (Placebo Comparator): no emitted particle at 20 bar pressure, identical in external appearance to Zingo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine (Zingo) — 0.5 mg lidocaine, 20 bar pressure
  Other Names: Zingo
  Arms: Lidocaine (Zingo)
Drug: Placebo — Placebo injector, 20 Bar pressure, empty injector
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of Zingo in treating pain associated with venipunture and peripheral venous cannulation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 3-12
* About to undergo venipuncture or peripheral venous cannulation at the back of the hand or antecubital fossa
* Have sufficient cognitive skills to identify faces depicting extremes of pain on the Wong-Baker FACES scale (age 3-12) and the extremes of pain on a 100 mm visual analog scale (VAS) (ages 8-12)
* Signed informed consent, cooperative and agree to attend follow-up visits

Exclusion Criteria:

* Any medical condition, non-compliance or instability (including but not limited to exceptionally upset, crying, anxiety) that in the judgement of the investigator might adversely affect the conduct of the study
* Used any (including external or inhaled) sedatives, analgesics, anaesthetics or other agents/device that may affect the efficacy assessment
* Subjects with tattoos, surgical scars, ports, implantable devices or a skin condition (e.g. excessive body hair) that may have interfered with the placement of Zingo or skin site assessments
* Active local infection or other skin pathology at the site of venipuncture or peripheral venous cannulation.
* Venipuncture of peripheral venous cannulation at the proposed site within the prior two weeks (longer if the wound is apparent)
* Previous history of allergic reactions to any local anaesthetic or tape/adhesive dressing.
* Participated in a clinical trial within three months prior to administration of study drug, or have already enrolled in a Zingo clinical trial before
* At the discretion of the investigator, any subjects that may have to be withdrawn from the study

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 288 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale After Venipuncture or Peripheral Cannulation | immediate after venipunture
  Child's assessment of pain on venipuncture or peripheral venous cannulation (all ages) performed one to three minutes after Zingo/Placebo administration, measured using the Wong-Baker FACES pain rating scale. The scale includes pictures of facial expressions with correlating numerical scale of 0-10, 0 being no hurt and 10 being the worst hurt.

SECONDARY OUTCOMES:
100-mm Visual Analogue Scale (VAS) | immediate after venipunture
  Assessment of pain on venipuncture or peripheral venous cannulation by children age 8-12, measured using a 100-mm VAS (0-100) anchored at 0 for "no pain" and at 100 for "worst possible pain."
Response Rate | immediate after venipunture
  Percentage of subject who score 0 or 1 in the FACES Pain Rating Scale
Compliance Score | immediate after venipunture
  Compliance to venipuncture assess by investigator

OTHER OUTCOMES:
Adverse Event Frequency | 1 day
Adverse Event Severity | 1 day
Comfort of Zingo/Placebo Administration (Wong-Baker) | immediate after venipunture
  Subject (all ages) to assess the level of comfort of Zingo/Placebo administration, measured using the Wong-Baker FACES scale (0-10), where 0 represent No Discomfort and 10 represent Worst Possible Discomfort.
Comfort of Zingo/Placebo Administration (VAS) | immediate after venipunture
  Subject (age 8-12) to assess the level of comfort of Zingo/Placebo administration, measured using VAS pain rating scales (0-100), where 0 represent No Discomfort and 100 represent Worst Possible Discomfort.
Local Adverse Reaction | Pre-dose (0-1 hour before), immediately after dose, 15 minutes, 30 minutes
  Local Adverse Reactions including erythema, edema, pruritus and hemorrhage/petechiae by severity.

CONTACTS AND LOCATIONS:
Overall Officials: Mazhong Zhang, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No